CLINICAL TRIAL: NCT04530565
Title: A Phase III Randomized Trial of Steroids + Tyrosine Kinase Inhibitor (TKI) Induction With Chemotherapy or Blinatumomab for Newly Diagnosed BCR-ABL-Positive Acute Lymphoblastic Leukemia (ALL) in Adults
Brief Title: Testing the Use of Steroids and Tyrosine Kinase Inhibitors With Blinatumomab or Chemotherapy for Newly Diagnosed BCR-ABL-Positive Acute Lymphoblastic Leukemia in Adults
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-06381; NCI-2020-06381 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA9181 (Other: ECOG-ACRIN Cancer Research Group); EA9181 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-08-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1
MeSH Terms: interventions — Specimen Handling; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Biopsy; Cyclophosphamide; Cytarabine; Dasatinib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Spinal Puncture; Mesna; Methotrexate; merphos; ponatinib; Prednisone; deltacortene; prednylidene; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (steroid, TKI), Single Arm Pre-Induction (Active Comparator): Patients receive prednisone PO QD on days 1-21 and ponatinib PO QD or dasatinib PO QD on days 1-21 based on investigator's choice.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Dasatinib; Procedure: Echocardiography Test; Procedure: Electrocardiography; Procedure: Lumbar Puncture; Procedure: Multigated Acquisition Scan; Drug: Ponatinib Hydrochloride; Drug: Prednisone
- Arm B (steroid, TKI, chemotherapy) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Electrocardiography; Procedure: Lumbar Puncture; Drug: Mesna; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Ponatinib Hydrochloride; Drug: Vincristine Sulfate
- Arm C (steroid, TKI, chemotherapy, immunotherapy) (Experimental): CYCLE 1: Patients receive ponatinib PO QD or dasatinib PO QD on days 1-28. Patients also receive dexamethasone PO or IV on day 1 and blinatumomab IV continuously on days 1-28, followed by methotrexate IT on day 29 or 30.
  CYCLE 2: Patients receive ponatinib PO QD or dasatinib PO QD on days 1-28. Patients also receive dexamethasone PO or IV on day 1 and blinatumomab IV continuously on days 1-28.
  Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Dasatinib; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: Electrocardiography; Procedure: Lumbar Puncture; Drug: Mesna; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Ponatinib Hydrochloride
- Arm D (steroid, TKI, chemotherapy, immunotherapy) (Experimental): Patients treated on Arm B who remain MRD positive at the end of induction therapy receive blinatumomab based re-induction identical to the regimen described for Arm C.
  Patients whose molecular test remains MRD positive after re-induction proceed to follow-up at the discretion of the investigator or receive anti CD-19 CAR- T cell therapy, inotuzumab ozogamicin, intensive chemotherapy, or palliative care.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cyclophosphamide; Drug: Dasatinib; Drug: Dexamethasone; Procedure: Echocardiography Test; Procedure: Electrocardiography; Procedure: Lumbar Puncture; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Ponatinib Hydrochloride
- Arm E (steroid, TKI, chemotherapy) (Experimental): Patients treated on Arm C who remain MRD positive at the end of induction therapy receive chemotherapy based re-induction which is identical to regimen described for Arm B according to patient's age and the pre-specified chemotherapy arm.
  Patients whose molecular test remains MRD positive after re-induction proceed to follow-up at the discretion of the investigator or receive anti CD-19 CAR- T cell therapy, inotuzumab ozogamicin, intensive chemotherapy, or palliative care.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Electrocardiography; Procedure: Lumbar Puncture; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Ponatinib Hydrochloride; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
  Arms: Arm C (steroid, TKI, chemotherapy, immunotherapy); Arm D (steroid, TKI, chemotherapy, immunotherapy)
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Arm B (steroid, TKI, chemotherapy); Arm D (steroid, TKI, chemotherapy, immunotherapy); Arm E (steroid, TKI, chemotherapy)
Drug: Cytarabine — Given IV or IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm B (steroid, TKI, chemotherapy); Arm E (steroid, TKI, chemotherapy)
Drug: Dasatinib — Given PO
  Other Names: BMS 354825; BMS-354825; BMS354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm B (steroid, TKI, chemotherapy); Arm C (steroid, TKI, chemotherapy, immunotherapy); Arm D (steroid, TKI, chemotherapy, immunotherapy); Arm E (steroid, TKI, chemotherapy)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
  Arms: Arm B (steroid, TKI, chemotherapy); Arm E (steroid, TKI, chemotherapy)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Electrocardiography — Undergo ECG
  Other Names: ECG; EKG
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Drug: Mesna — Given IV
  Other Names: 2-Mercaptoethanesulfonate, Sodium Salt; Ausobronc; D-7093; Filesna; Mercaptoethane Sulfonate; Mercaptoethanesulfonate; Mesnex; Mesnil; Mesnum; Mexan; Mistabron; Mistabronco; Mitexan; Mucofluid; Mucolene; UCB 3983; Uromitexan; Ziken
  Arms: Arm B (steroid, TKI, chemotherapy); Arm C (steroid, TKI, chemotherapy, immunotherapy)
Drug: Methotrexate — Given IV or IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm B (steroid, TKI, chemotherapy); Arm C (steroid, TKI, chemotherapy, immunotherapy); Arm D (steroid, TKI, chemotherapy, immunotherapy); Arm E (steroid, TKI, chemotherapy)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; MUGA; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Ponatinib Hydrochloride — Given PO
  Other Names: AP24534 HCl; Iclusig
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm A (steroid, TKI), Single Arm Pre-Induction
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm B (steroid, TKI, chemotherapy); Arm E (steroid, TKI, chemotherapy)

SUMMARY:
This phase III trial compares the effect of usual treatment of chemotherapy and steroids and a tyrosine kinase inhibitor (TKI) to the same treatment plus blinatumomab. Blinatumomab is a Bi-specific T-Cell Engager ('BiTE') that may interfere with the ability of cancer cells to grow and spread. The information gained from this study may help researchers determine if combination therapy with steroids, TKIs, and blinatumomab work better than the standard of care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the overall survival (OS) following induction with steroids + TKI + blinatumomab versus induction with steroids + TKI + chemotherapy.

SECONDARY OBJECTIVES:

I. To compare the rate of minimal residual disease (MRD) negativity for patients treated with chemotherapy versus (vs) blinatumomab at the end of first induction (week 15).

II. To evaluate the rate of the MRD negativity by treatment arm for those patients MRD positive after the first induction and administered of second induction.

III. To compare event free survival (EFS) for patients initially randomized for chemotherapy vs blinatumomab.

IV. To assess the toxicities of blinatumomab + TKI vs. TKI + chemotherapy in this patient population.

V. To assess the toxicities of the chemotherapy regimen in this patient population.

VI. To describe the outcome of patients who proceed to allogeneic stem cell transplant after treatment with blinatumomab + TKI only.

OUTLINE:

ARM A (PRE-INDUCTION): Patients receive prednisone orally (PO) once daily (QD) on days 1-21 and ponatinib hydrochloride (ponatinib) PO QD or dasatinib PO QD on days 1-21 based on investigator's choice.

Patients are randomized to 1 of 2 arms (Arm B or C). Patients undergo bone marrow aspiration with biopsy, lumbar punctures, echocardiogram (ECHO), and multigated acquisition (MUGA) scans as indicated by investigator.

ARM B (INDUCTION THERAPY):

CYCLE 1: Patients receive cyclophosphamide intravenously (IV) twice daily (BID) on days 1-3, dexamethasone PO or IV on days 1-4 and 11-14, cytarabine intrathecally (IT) on day 1, doxorubicin hydrochloride (doxorubicin) IV on day 4, vincristine sulfate (vincristine) IV on days 4 and 11, and methotrexate IT on day 8. Patients also receive Mesna 600mg/m^2 IV as a 'chemoprotectant' via continuous infusion on days 1-3, (beginning 1 hour prior to cyclophosphamide and completed by 12 hours after the last dose of cyclophosphamide).

CYCLE 2 (AGE 18-70): Starting in cycle 2, fit patients aged 18-70 receive dasatinib 70mg/day PO QD or ponatinib 30mg/day PO QD on days 1-21, methotrexate IV over 24 hours and IT on day 1, and cytarabine IV over 2 hours BID on days 2-3 of each cycle. On day 22 of cycle 2 or later, as soon as the absolute neutrophil count (ANC) is greater than 1000 cells/ul and platelets are greater than 50,000 cells/ul, patients receive hyper cyclophosphamide, vincristine, doxorubicin, and dexamethasone (CVAD) for 2 additional cycles.

CYCLE 2 (AGE > 70 or unfit < 70): Starting in cycle 2, patients age > 70 or younger unfit patients for Hyper-CVAD receive ponatinib PO QD or dasatinib PO QD on days 1-21 of each cycle. Patients also receive methotrexate IV over 24 hours and IT on day 1, and cytarabine IV over 2 hours BID on days 2-3 of each cycle. Cycle 1 and 2 regimens are each repeated once starting on day 22 of cycle 2, or later, but as soon as the ANC is greater than 1000 cells/ul and platelets are greater than 50,000 cells/ul.

Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve remission (significant reduction in the amount of leukemia in bone marrow and blood/MRD negative) after 4 cycles may receive alternative treatment, either consolidation with two cycles of Hyper-CVAD followed by TKI maintenance therapy or undergo allogeneic stem cell transplantation followed by maintenance therapy. Patients who do not achieve a remission (MRD positive) are assigned to Arm D. Patients who experience un-resolving renal failure or life-threatening infection which may require a treatment delay of 21 days cross-over to Arm C to receive the prescribed course of blinatumomab.

ARM C (INDUCTION THERAPY):

CYCLE 1: Patients receive ponatinib PO QD or dasatinib PO QD on days 1-28. Patients also receive dexamethasone PO or IV on day 1 and blinatumomab IV continuously on days 1-28, followed by methotrexate IT on day 29 or 30.

CYCLE 2: Patients receive ponatinib PO QD or dasatinib PO QD on days 1-28. Patients also receive dexamethasone PO or IV on day 1 and blinatumomab IV continuously on days 1-28.

Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

ARM D (RE-INDUCTION): Patients treated on Arm B who remain MRD positive at the end of induction therapy receive blinatumomab based re-induction identical to the regimen described for Arm C.

ARM E (RE-INDUCTION): Patients treated on Arm C who remain MRD positive at the end of induction therapy receive chemotherapy based re-induction which is identical to regimen described for Arm B according to patient's age and the pre-specified chemotherapy arm.

Patients whose molecular test remains MRD positive after re-induction proceed to follow-up at the discretion of the investigator or receive anti CD-19 CAR- T cell therapy, inotuzumab ozogamicin, intensive chemotherapy, or palliative care.

Patients are followed up every 3 months for first 2 years (from study registration), every 6 months for years 3-5, and then every 12 months for years 6-10.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA FOR PRE-REGISTRATION (TO STEP 0)
* Patient must be >= 18 and =< 75 years of age
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status between 0-3
* Patient must be newly diagnosed with B acute lymphoblastic leukemia (B-ALL) or is suspected to have acute lymphoblastic leukemia (ALL)

  * Patient must have BCR-ABL1 positive disease. The diagnosis of ALL and the presence of BCR-ABL translocation must be confirmed centrally. Patients can be registered and begin step 1 therapy while awaiting central laboratory eligibility confirmation

    * NOTE: Bone marrow aspirate and/or peripheral blood specimen must be submitted to the ECOG-American College of Radiology Imaging Network (ACRIN) Leukemia Laboratory at MD Anderson Cancer Center to determine patient's eligibility for registration to Step 1 or confirm patient evaluability. Centrally fluorescence-activated cell sorting (FACS) analysis will be performed to determine B-ALL and to exclude acute myeloid leukemia (AML) or acute bi-phenotypic leukemia and baseline BCR-ABL status will be determined by fluorescent in situ hybridization (FISH). The ECOG-ACRIN Leukemia Laboratory will forward results within 48 hours of receipt of the specimen to the submitting institution. Bone marrow aspirate is to be from first pull (initial or re-direct). Specimens must contain sufficient blast cells. In cases where the bone marrow aspiration may be inadequate, or the bone marrow examination has already been performed prior to study consent and enrollment on Step 0, peripheral blood may be submitted, with recommendation that adequate circulating blasts are present (> 10%). If a diagnosis of BCR-ABL positive B-ALL has already been established by local Clinical Laboratory Improvement Act (CLIA) certified laboratories, the patient may be registered to step 1 without waiting for central confirmation
* Patient must not have a diagnosis of BCR/ABL T-ALL
* Patient must not have received chemotherapy for B-ALL. Patients who received up to five days of therapy (hydroxyurea and/or steroids of any kind) with the aim to reduce disease burden prior to study registration to Step 1 are eligible
* Patient must not have unstable epilepsy that requires treatment
* Patients with lymphoid blast crisis chronic myeloid leukemia (CML) are not eligible
* ELIGIBILITY CRITERIA FOR REGISTRATION TO STEP 1
* Patient must have a diagnosis of Philadelphia chromosome positive (Ph+) ALL that has been determined locally and bone marrow and/or peripheral blood was sent and receipt confirmed for central confirmation or determined centrally by the ECOG-ACRIN Leukemia Laboratory at MD Anderson Cancer Center
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy. A patient of childbearing potential is defined as any woman, regardless of whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse from the time of step 1 registration, while on study treatment, and until at least six months after the last dose of study treatment
* Total bilirubin =< 3 mg/dL (patients with Gilbert's syndrome must have a total bilirubin =< 5 mg/dL) (obtained =< 28 days prior to step 1 registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X the institutional upper limit of normal (ULN) (obtained =< 28 days prior to step 1 registration)
* Estimated creatinine clearance > 45 mL/min (based on Cockcroft-Gault equation) (obtained =< 28 days prior to step 1 registration)
* Patients with acute organ dysfunction at step 1 registration, which may be attributed to leukemia can be registered regardless of lab results at presentation. Such patients will be allowed to register and can start Arm A steroid + TKI therapy but will only be allowed to proceed to step 2 randomization if the eligibility criteria outlined is met
* Patients who presented with no evidence of acute organ dysfunction but during step 0 experienced a rise in liver enzymes which investigator suspects to be a side effect of any of prescribed drugs, are allowed to be registered regardless of the level of liver enzymes. Step 2 randomization must be withheld until the eligibility criteria outline is met but no more than 14 days after concluding Arm A therapy
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable or on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have an undetectable HCV viral load and if indicated, on treatment
* Patients with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must not have active concomitant malignancy. Patients on chronic hormonal therapy for breast or prostate cancer or patients treated with maintenance with targeted agents but are in remission with no evidence for the primary malignancies are eligible
* Patient must not have complaints of symptoms and/or have clinical and/or radiological signs that indicate an uncontrolled infection or any other concurrent medical condition that could be exacerbated by the treatment or would seriously complicate compliance with the protocol
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients must be class 2B or better
* Investigators must confirm which TKI patient is to receive

  * NOTE: Patients with known T315I mutation status should receive ponatinib treatment
  * NOTE: In situations due to insurance coverage issues and the pre-selected TKI is not immediately available, patients can receive dasatinib or imatinib during step 1. The investigator must re-specify dasatinib or ponatinib prior to step 2 randomization and from then on patients must receive the pre-selected TKI only
* ELIGIBILITY CRITERIA FOR RANDOMIZATION TO STEP 2
* Patient must have completed at least 7 and no more than 21 days of protocol-treatment on Arm A prior to step 2 randomization. (Days in which arm A therapy was withheld for any reason are not counted)

  * NOTE: First day of steroids prescription after registration will be considered as the first day of study therapy. The selected TKI must be initiated prior to randomization
* Patients who presented with acute organ dysfunction within 2 weeks of registration to step 1 must have total bilirubin =< 2 X institutional upper limit of normal (ULN)
* AST(SGOT) and ALT(SGPT) =< 2 X the institutional upper limit of normal (ULN)
* Estimated creatinine clearance > 45 mL/min (based on Cockcroft-Gault equation)
* Investigators must confirm which TKI patient is to receive.

  * NOTE: Patients with known T315I mutation status should receive ponatinib treatment
* For patients under age 70, intended chemotherapy regimen must have been determined prior to randomization
* Patient must not have active central nervous system (CNS) involvement by leukemic blasts. Patients with signs of CNS involvement at presentation are eligible for randomization if clearance of blasts from the cerebrospinal fluid (CSF) is demonstrated
* Patients must have resolved any serious infectious complications related to therapy
* Any significant medical complications related to therapy must have resolved
* ELIGIBILITY CRITERIA FOR REGISTRATION TO STEP 3 (RE-INDUCTION)
* Institution has received centralized MRD results confirming positive status
* Patients who presented with acute organ dysfunction within 2 weeks of registration to step 1 must have total bilirubin =< 2 X institutional ULN
* Patients who presented with acute organ dysfunction must have AST (SGOT)/ALT (SGPT) =< 2 X institutional upper limit of normal (ULN)
* Patients who presented with acute organ dysfunction must have an estimated creatinine clearance > 45 mL/min (based on Cockcroft-Gault equation)
* Investigators must confirm which TKI patient is to receive

  * NOTE: Patients with known T315I mutation status should receive ponatinib treatment
* For patients under age 70 and previously assigned to Arm C, intended chemotherapy regimen must have been determined
* Step 3 (Re-Induction): Patients must have resolved any serious infectious complications related to therapy
* Step 3 (Re-Induction): Any significant medical complications related to therapy must have resolved

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Time between randomization and death from any cause, assessed up to 10 years from the date of registration
  Will compare OS following induction with steroids + tyrosine kinase inhibitor (TKI) + blinatumomab and induction with steroids + TKI + chemotherapy. Will be based on an intent-to-treat analysis. Estimates of OS including medians and confidence intervals, will be calculated using the Kaplan-Meier method. Comparisons of OS between treatment arms will be conducted using the one-sided stratified log-rank test with steroid responsiveness, type of TKI intended to receive and age at diagnosis, the same factors used in randomization, as stratification factors. Cox proportional hazards models of OS, stratified on the same factors used in the randomization, will be used to assess the effect of treatment by adjusting other possible clinical and biological risk factors, including cytogenetic abnormalities.

SECONDARY OUTCOMES:
Rate of minimal residual disease (MRD) negativity | At week 15
  Will be centrally evaluated. Will be compared between two arms using Fisher's exact test with a one-sided type I error rate of 2.5%. Multivariable logistic regression modeling will be used to adjust for other possible clinical and biological risk factors. For patients registered to Step 3 (re-induction), the rates of MRD negativity and their corresponding 95% confidence intervals after re-induction will be given by treatment arm.
Event free survival (EFS) | Time from randomization to failure to achieve induction molecular remission by week 15, confirmed molecular relapse after molecular remission or to death in remission, assessed up to 10 years from the date of registration
  Will be based on an intent-to-treat analysis. Estimates of EFS including medians and confidence intervals, will be calculated using the Kaplan-Meier method. Comparisons of EFS between treatment arms will be conducted using the one-sided stratified log-rank test with steroid responsiveness, type of TKI intended to receive and age at diagnosis, the same factors used in randomization, as stratification factors. Cox proportional hazards models of EFS, stratified on the same factors used in the randomization, will be used to assess the effect of treatment by adjusting other possible clinical and biological risk factors, including cytogenetic abnormalities
Rate of MRD negativity | After re-induction
  Will be centrally evaluated. Will be compared between two arms using Fisher's exact test with a one-sided type I error rate of 2.5%. Multivariable logistic regression modeling will be used to adjust for other possible clinical and biological risk factors. For patients registered to Step 3 (re-induction), the rates of MRD negativity and their corresponding 95% confidence intervals after re-induction will be given by treatment arm.
Incidence of adverse events | Up to 10 years from the date of registration
  All toxicity grades and reportable adverse events will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yishai Ofran, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (211):
- United States (207):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Yale University, New Haven, Connecticut
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm